CLINICAL TRIAL: NCT03861182
Title: Contribution of PRF (Platelet Rich Fibrin) in the Biological Functionalization of Prothetic Patch Closure : in Vitro Study
Brief Title: Contribution of PRF in CDH in Children With Prothetic Patch Closure
Acronym: HECODIAP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of staff
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 7067
Record Dates: First submitted 2019-01-24; First posted 2019-03-04 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2019-09

CONDITIONS: Congenital Diaphragmatic Hernias
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adult Healthy Volunteers (Other)
  Interventions: Biological: Biological functionalization of the prosthetic materials by PRF
- Neonates (Other)
  Interventions: Biological: Biological functionalization of the prosthetic materials by PRF

INTERVENTIONS:
Biological: Biological functionalization of the prosthetic materials by PRF — The biological functionalization of the prosthetic materials by host PRF would improve the biological colonization of materials and thus reduce the risk of prosthetic release.

SUMMARY:
Improved management of giant congenital diaphragmatic hernias (CDH) in neonates : decreased risk of morbidity and mortality due to prosthesis release. CDH is a rare disease with a still very dark prognosis, with a high rate of morbidity and mortality in giants forms linked to the release of insufficiently biologically integrated prosthesis. The biological functionalization of the prosthetic materials by host PRF would improve the biological colonization of materials and thus reduce the risk of prosthetic release.

ELIGIBILITY:
Inclusion Criteria:

Adult Healthy Volunteers :

- Over 18 years of age

Neonates:

* Aged between 1h of life and 28 days of life
* Born beyond 33 Week of Amenorrhea + 1day and 2kg of birth weight
* Hospitalized in the medical-surgical centre of Pediatrics of the hospital of Strasbourg
* For whom a blood sample was prescribed as part of their routine care

Exclusion Criteria:

Adult Healthy Volunteers :

* Systemic inflammatory disease
* Transient inflammatory state
* Any drug that modifies the coagulation cascade during the 48h preceding the sampling

Neonates:

* Risk of anemia < 7g/DL
* Current anticoagulant treatment

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Comparison of cell colonization between neonate biomaterials and the same biomaterials functionalized by Platelet Rich Fibrin of healthy adult volunteers. | 7 days
  Analysis of cell colonization after cell culture.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France